CLINICAL TRIAL: NCT04009993
Title: A-BIRTHPERFORM Versus Conventional Partogram in the Improvement of Birth Results: a Randomized Controlled Trial
Brief Title: A-BIRTHPERFORM Versus Conventional Partogram in the Improvement of Birth Results
Acronym: A-BRTHPRFORM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, LAURA GARCIA-LAUSIN, Principal Investigator, Hospital del Mar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SLT0 06/17/0 0 011
Record Dates: First submitted 2019-05-06; First posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Labor Complication
Keywords: digital tool; decision making; labour process; birth results
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-BIRTHPERFORM digital tool (Experimental): interactive partogram that maternity care professionals of the experimental group use, in interactive and device will guide the professional thought the NICE guidelines on labour care
  Interventions: Device: A-BIRTHPERFORM digital tool
- control group with conventional partogram use (No Intervention): Conventional care in each participant hospital, with conventional partogram in each centre

INTERVENTIONS:
Device: A-BIRTHPERFORM digital tool — use of A-BIRTHPERFORM digital tool
  Arms: A-BIRTHPERFORM digital tool

SUMMARY:
Midwives and Obstetricians when assisting women during labour do not follow the clinical guidelines on labour process care,in many cases oxytocin is used routinely without medical indication, and ends in the erroneous use of oxytocin, and risk of labour dystocia arise. In Spain, according to the National Health System the rate of oxytocin use during labour is 53.3%, in pregnant women with spontaneous onset of labour, which is high and is far from the expected standard (expected standard of 5 to 10%, as an indicator of good practice). The partogram is one of the conventional obstetric tools used in labour wards, specially the World Health Organization partogram with the four-hours action line, which is widely used and it serves to give a graphic content and a global vision of the evolution and medication given in a concrete women in labour, although a routine use of partogram is not recommended, and new studies are needed to stablish the effectiveness of the partograph. There are frequent professional errors using conventional partogram and this justify the need for a tool different from the usual ones. The algorithm of care in normal and in disrupted labour recommended by The National Institute for Health and Clinical Excellence (NICE) guidelines is complex.

The tool the investigators have designed is A-BIRTHPERFORM digital tool for professionals and consists in helping applying the Intrapartum Care´s NICE Guidelines algorithms to help decision-making.

Objective: The aim of the study will be to analyze if the use of A-BIRTHPERFORM contributes to improve perinatal results by reducing instrumental deliveries and caesarean sections.

Methods: Design: randomized controlled trial. Participants: The study will be conducted in 4 maternity hospitals of different autonomous communities of Spanish. Participants will be women from 18 to 41 years of age, pregnant at term between 37 and 41 weeks gestation, with spontaneous onset of labour or induced labour and with low or medium obstetric risk. Participants will be randomized to receive professional care during delivery using A-BIRTHPERFORM or assigned to conventional partogram care. The control group will be subject to traditional care through the use of conventional partogram used in each hospital following the labour care guidelines of each participant hospital. The experimental group will be cared by professionals using A-BIRTHPERFORM during the whole labour process.

Discussion: A-BIRTHPERFORM could help improve the use of NICE Guidelines on Intrapartum Care, and could help reducing the use of oxytocin, decreasing instrumented deliveries and severe perineal lacerations. The digital tool aims to provide standardization and systematization to childbirth care and to serve as a communication tool between team members.

This tool could allow the professional to freely access it from any digital device, not necessarily located at the counter or reception of the maternal unit, which facilitates personal reflection on labour progress and with the team, in order to improve health results for women and their families.

DETAILED DESCRIPTION:
Stimulation of labour with synthetic oxytocin is increasingly used all over the world. Synthetic oxytocin is used in cases of dystocia of labour, with the objective of attempting labour progression until achieving vaginal birth. The use of oxytocin could have potential adverse effects on the mother and the fetus, such as uterine tachysystole, which can lead to uterine rupture and fetal distress . There is a risk of fetal hypoxemia and acidemia if the contractions are very frequent and prolonged. The risk of instrumented delivery is even higher when oxytocin is used when labour is progressing normally. There is a significant association between oxytocin use to stimulate labour and severe perineal lacerations, postpartum urinary retention, postpartum hemorrhage and delayed onset of breastfeeding. The World Health Organization (WHO) defines dystocia of labour as four hours without progress during the active labor and is recommended to medically intervene . When health professionals that assist women in labour (Midwives and Obstetricians) do not follow the clinical guidelines on intrapartum care, labour dystocia and oxytocin use, and oxytocin is used routinely without medical indication, ends in the erroneous use of oxytocin. According to the evaluation of Strategy of Attention to Normal Childbirth (SANC), the National Health System in Spain, which sets standards of quality in obstetric practice, showed a rate of 53.3% of oxytocin use during labor in pregnant women with spontaneous onset of labour, which is high and is far from the expected standard (expected standard of 5 to 10%, as an indicator of good practice).

According to the Romano and de Lothian study, a high use of oxytocin during labour would be related to the so-called "cascade of interventions", referring to different obstetric interventions that are used routinely and not based on scientific evidence which could interfere in the physiology of childbirth and in the skills of women to cope with labour and labour pain. The use of oxytocin has a limited and uncertain benefit , and may even be harmful in some specific situations during labor. Lothian suggests in his study that routine practices that are unnecessary in physiological births should be avoided, thus minimizing complications, and improving perinatal outcomes.

An international consensus was published in 2017 to review the scientific evidence on care practices that facilitate a physiological delivery process and its relationship with the improvement of perinatal outcomes and maternal satisfaction.

The increase in the use of oxytocin during childbirth in healthy women and with spontaneous onset of labour seems to be generalized worldwide, and national and international agencies demand an improvement in the care provided during childbirth in women with pregnancies of low obstetric risk, with the objective of limiting unnecessary interventions during childbirth and birth.

In the same line, in 2018 an international initiative for childbirth (ICI) is promoted with 12 steps towards a safe and respectful Mother-Family motherhood, ICI-Mother Baby Childbirth Organization (IMBCO) and International Federation of Gynecology and Obstetrics (FIGO), in which "step 6" recommends: Promote and provide clinical practice based on evidence that has proven to be beneficial and respect the normal physiology of labour. Allowing labour to develop at its own pace, avoiding unnecessary interventions.

In Spain, although the guidelines on Normal Childbirth recommends not to perfuse oxytocin routinely during labour, since the evidence shows that this does not improve the results (SANC), the rate of 53% of oxytocin shows that it seems to be routinely used. Routine oxytocin use´s consequences are: increase in cesarean and instrumental deliveries, loss of fetal wellbeing intrapartum, uterine rupture, among others.

The partogram is one of the conventional obstetric tools used in labour wards, specially the World Health Organization partogram with the four-hours action line, which is widely used and it serves to give a graphic content and a global vision of the evolution and medication given in a concrete women in labour, although a routine use of partogram is not recommended, and new studies are needed to stablish the effectiveness of the partogram. There are frequent professional errors using conventional partogram and this justify the need for a tool different from the usual ones. The algorithms of care in normal and in disrupted labour care of The National Institute for Health and Clinical Excellence guidelines are complex. The use of a tool for professionals that facilitate decision making by following the clinical practice guidelines could ensure the guidelines are followed-up properly and improve quality of care, patients safety related aspects and improve the results of childbirth for women and the neonates.

The tool the investigators are developing is called A-BIRTHPERFORM and consists of the clinical guidelines algorithms to help decision-making based on scientific evidence. The algorithm takes into account the specific labour phase and the women characteristics ( first or second stage of labour, and if in second stage of labour the algorithm differentiate if latent or active phase of this stage), the parity (nulliparous or multiparous women) and shakes into account whether the women uses epidural analgesia as pain relief during labour. It would be like an interactive partogram, where the professional will be guided through the appropriate algorithm of care during the labour process. There is evidence about the use of digital tools for professionals in different areas of health. In the area of maternity care the investigators have found evidence on digital tools for cardiotocographic interpretation, or as an aid for health professional for decision making on women admission to labour ward. The investigators have not found any evidence about this type of tool proposed, for its specific intrapartum care use. It seems to be a lack of research studies on digital tools in childbirth providing clinical and therapeutic advantages in birth results in relation to pre-technological care.

A-BIRTHPERFORM could help reduce the use of oxytocin, decrease instrumented deliveries and severe perineal lacerations that seem to be directly related to the use of oxytocin . The digital tool aims to provide standardization and systematization to childbirth care and to serve as a communication tool between team members. Digital tools for health professionals have proven to be effective to support a better decision making and better results in patients and users of health services.

For the development of A-BIRTHPERFORM digital tool the investigators are been supported by Hospital del Mar Medical Research Institute (IMIM). A-BIRTHPERFORM will be tested to evaluate its comprehensibility, acceptability and viability. This tool aims to be an aid for clinicians, both in the monitoring and support during normal birth, and in complex situations helping to determine at each moment of the process how to intervene during labour, in case of labour dystocia for example, by artificially rupturing the membranes or by using oxytocin, or for arrested labour by performing an instrumented delivery or cesarean section.

On the other hand, this tool allows the professional to freely access from any digital device, not necessarily located at the counter or reception of the maternal unit, which facilitates personal reflection on labour progress and with the team, in order to improve health results for women and their families.

The purpose of the investigators is to assess whether A-BIRTHPERFORM improves perinatal outcomes compared with conventional partogram use.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age: 37-41 weeks
* Spontaneous and induced onset of labour
* Women with low and medium risk during labour and birth with cephalic presentation fetus

Exclusion Criteria:

* Premature
* High risk pregnancies and labour
* Malpositions of the fetus

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 969 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of non-spontaneous vaginal births | Immediately after the birth
  Investigator will be making this evaluation after birth, evaluating the data obtained from the conventional partogram (in the control group) and from the A-BIRTHPERFORM tool (in the intervention group). The measurements or variables that will be used are: data of the progress of labour entered against time, cervical dilatation, record of start oxytocin use if necessary, time of birth, and birth mode in each group of the trial

SECONDARY OUTCOMES:
Percentage of compliance with NICE clinical guidelines on artificial rupture of membranes technique | Immediately after the birth
  Investigator will be making this evaluation after birth, evaluating the data obtained from the conventional partogram (in the control group) and from the A-BIRTHPERFORM tool (in the intervention group). The measurements that will be used are birth progress variables/ parameters: data of the progress of labour entered against time, cervical dilatation, record of time artificial rupture of membranes perform variable. Investigator will assess compliance of NICE clinical guidelines on active labour, that states that if progress of cervical dilatation in four hour's time is less than 2cm of cervical dilatation an artificial rupture of membranes should be performed to help with the progress of labour.
  Investigators will be comparing compliance of guidelines on artificial rupture of membranes between control group and intervention group and evaluating the percentage of compliance of this technique following the guidelines.
Percentage of compliance with NICE clinical guidelines on oxytocin use during labour | Immediately after the birth
  Investigator will be making this evaluation after birth, evaluating the data obtained from the conventional partogram (in the control group) and from the A-BIRTHPERFORM tool (in the intervention group). The measurements or variables that will be used are: data of the progress of labour entered against time, cervical dilatation, and oxytocin use variable. Investigator will assess compliance of NICE clinical guidelines on active labour that states that in case of spontaneous rupture of membranes if progress is less than 2cm of cervical dilatation in four hours NICE clinical guidelines recommends starting use of oxytocin, or in case or artificial rupture of membranes when the progress is less than 1cm of cervical dilatation in two hours, form the data collected conventional partogram (in the control group) and from the A-BIRTHPERFORM tool (in the intervention group) investigators will analyze the trial´s participants following the guidelines.

IPD SHARING:
Plan to Share IPD: No